CLINICAL TRIAL: NCT05932485
Title: Effect of Stellate Ganglion Block on New Atrial Fibrillation After Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, MD, the Deputy Director of Anesthesiology, the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20230609
Record Dates: First submitted 2023-06-10; First posted 2023-07-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stellate Ganglion Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left stellate ganglion block (Experimental): Left stellate ganglion block under ultrasound guidance was administered with 0.375% Ropivacaine hydrochloride 5 ml
  Interventions: Procedure: Stellate nerve block
- Control (No Intervention): do nothing

INTERVENTIONS:
Procedure: Stellate nerve block — Before the operation, the left stellate ganglion block was performed, and 0.375% ropivacaine 5ml was injected into the stellate ganglion.
  Arms: Left stellate ganglion block

SUMMARY:
Post-operative new-onset atrial fibrillation (POAF) is one of the most common arrhythmias in adults after direct intracardiac surgery with extracorporeal circulation. The incidence of POAF in coronary artery bypass grafting (CABG) is approximately 30%. POAF can lead to an increased risk of complications such as stroke, heart failure, and acute kidney injury, which not only prolongs the patient's hospital stay, but also increases hospital costs and mortality. operation, extracorporeal circulation, and the patient's underlying conditions (such as age, gender, hypertension, and diabetes), which cause sympathetic activation, inflammatory response, and myocardial ischemia in the organism. The stellate ganglion block (SGB) regulates the sympathetic tone of the innervated nerves and thus the autonomic function of the body. SGB can effectively regulate the sympathetic-parasympathetic imbalance. Also, SGB may exert some anti-inflammatory effects. In this study, ultrasound-guided SGB was used in CABG patients to investigate its effect on the occurrence of POAF.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first-time and elective coronary artery bypass grafting;
* ASA grade II-IV；
* The preoperative ECG showed sinus heart rate.

Exclusion Criteria:

* The patient refused to participate in this study;
* Surgical procedures include any other type of heart surgery in addition to CABG；
* Allergic to known general anesthesia drugs;
* Patients with a history of neck surgery or abnormal neck anatomy;
* Patients with contraindications to SGB.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of new atrial fibrillation was detected by ECG monitoring | Within 5 days after surgery
  ECG monitor shows atrial fibrillation. To be specific: 1)Irregular R-R interval (when atrioventricular conduction is present), 2) P wave disappearance, 3) irregular atrial activity.

SECONDARY OUTCOMES:
AF burden | within 5 days after surgery
  The percentage of the time during which atrial fibrillation occurs in the overall recorded time.
Duration of the first episode of POAF | within 5 days after surgery
  The duration from the onset to the resolution of the first atrial fibrillation after surgery.
Need for Antiarrhythmic treatments | within 5 days after the operation
  Record the types of medications used and whether electrical cardioversion has been used.
the concentration of interleukin-6 | end of surgery, 24 hour postoperatively, 72hour postoperatively, 5 day postoperatively
  Interleukin-6 (IL-6) is an important cytokine that plays a key role in immune responses, inflammation, and tumor development.
the concentration of CRP | end of surgery,24 hour postoperatively ,72 hour postoperatively ,5 day postoperatively
  C-reactive protein (CRP) is a protein produced by the liver that is mainly used to indicate the presence of inflammation in the body.
Changes of intraoperative Left ventricular diastolic function | T1 (after sternotomy and before CPB) and T2 (30 minute after CPB cessation).
  Left ventricular diastolic function were measured by transesophageal echocardiography (TEE)
the concentration of Hs-cTnT | end of surgery, 24hour postoperatively, 72hour postoperatively
  hs-cTnT is an important biomarker used for detecting cardiac injury.
the concentration of CK-MB | end of surgery, 24hour postoperatively, 72hour postoperatively
  CK-MB is an enzyme primarily found in cardiac muscle cells. Its concentration is commonly used to assess cardiac damage, especially in the case of myocardial infarction
postoperative adverse reactions | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Record the occurrence of adverse reactions postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China